CLINICAL TRIAL: NCT07320001
Title: Injection Sclerotherapy With Bleomycin VS Doxycycline in Patients With Lymphatic Malformations:A Randomized Controlled Trial
Brief Title: Injection Sclerotherapy With Bleomycin VS Doxycycline in Patients With Lymphatic Malformations
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Basharat Hussain (Other)
Responsible Party: Sponsor-Investigator, Basharat Hussain, Principal Investigator, Holy Family Hospital, Pakistan
Organization: Holy Family Hospital, Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-RCT-01
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Lymphatic Abnormality
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Bleomycin; Doxycycline; Tetracycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bleomycin sclerotherapy (Active Comparator)
  Interventions: Drug: Bleomycin
- Doxycycline sclerotherapy (Experimental)
  Interventions: Drug: doxycycline (tetracycline)

INTERVENTIONS:
Drug: Bleomycin — Injection sclerotherapy using bleomycin administered according to standard hospital protocol. The number of sessions and dosage are determined based on lesion size and patient response. Safety and adverse events are monitored by the principal investigator and treating physicians.
  Arms: Bleomycin sclerotherapy
Drug: doxycycline (tetracycline) — Injection sclerotherapy using doxycycline administered according to hospital protocol. The number of sessions and dosage are determined based on lesion size and patient response. Safety and adverse events are monitored by the principal investigator and treating physicians.
  Arms: Doxycycline sclerotherapy

SUMMARY:
This is a randomized clinical trial comparing the safety and effectiveness of injection sclerotherapy using bleomycin versus doxycycline in children under 12 years with lymphatic malformations. The study will assess reduction in lesion size, clinical improvement, and treatment-related complications over six months.

DETAILED DESCRIPTION:
This randomized clinical trial aims to compare the effectiveness and safety of injection sclerotherapy using bleomycin versus doxycycline in pediatric patients under 12 years of age diagnosed with lymphatic malformations. Eligible participants will be randomly assigned to receive either bleomycin or doxycycline injections at Holy family hospital Rawalpindi Pakistan.

The study will monitor participants over a six-month follow-up period to assess primary outcomes, including reduction in lesion size and clinical improvement, as well as secondary outcomes such as treatment-related complications, number of treatment sessions required, and overall patient tolerance.

Standard hospital protocols for injection sclerotherapy will be followed, and safety will be monitored by the principal investigator and treating physicians. Participants' caregivers will provide informed consent prior to enrollment. This study is designed to provide evidence on the comparative effectiveness of bleomycin versus doxycycline for pediatric lymphatic malformations

ELIGIBILITY:
Inclusion Criteria:

Age 0-12 years Radiological diagnosis of macrocytic/mixed lymphatic malformations. No prior sclerotherapy/surgical treatment. Informed consent from guardians

-

Exclusion Criteria:

* microcytic lymphatic malformations Allergies to bleomycin/Doxycycline. Significant co morbidities Active infection at lesion site.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Change in lymphatic malformation volume from baseline at 6 months | 6 months.
  Change in lymphatic malformation size measured as percentage reduction in lesion volume from baseline, assessed using ultrasonography (or MRI, if you are using MRI) at baseline and at 6 months after sclerotherapy.

SECONDARY OUTCOMES:
Number of participants with treatment-related complications within 6 months | 6 months.
  Number of participants who develop treatment-related complications, including pain, fever, infection, skin necrosis, swelling, or ulceration, assessed clinically and graded using CTCAE v5.0 (or v4.0) within 6 months after sclerotherapy.